CLINICAL TRIAL: NCT01405274
Title: Exploring the Impact of a Physiotherapy Intervention on the Risk of Re-injury and Recovery in Children and Adolescents With Acute Ankle Sprains: a Randomized Controlled Trial
Brief Title: Impact of Physiotherapy Intervention for Children With Ankle Sprains
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Principal Investigator, Isabelle Gagnon, Clinical Scientist, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 09-287-PED
Record Dates: First submitted 2011-07-28; First posted 2011-07-29 (Estimated); Last update posted 2019-04-04 (Actual); Status verified 2019-04

CONDITIONS: Physical Therapy
MeSH Terms: interventions — Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Physiotherapy intervention (Experimental)
  Interventions: Other: Physiotherapy
- standard care (No Intervention)

INTERVENTIONS:
Other: Physiotherapy — Physiotherapy treatment bi-weekly, delivered at the child's home
  Arms: Physiotherapy intervention

SUMMARY:
This study will investigate whether adding a physiotherapy intervention to standard Emergency Department care will lead to improved recovery following an ankle sprain in the pediatric and adolescent population as well as to a decrease recurrence of injuries during the year following the initial ankle sprain. Children will be allocated to standard care or to the added intervention group. The study hypothesis is that recovery will be better while recurrence of injury will be less in those receiving the added physiotherapy intervention.

ELIGIBILITY:
Inclusion Criteria:

* age 7 to 18
* confirmed diagnosis of ankle sprain
* Ability to Speak French or English

Exclusion Criteria:

* immobilization at the time of ED discharge

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 170 (Actual)
Dates: Start 2011-07; Primary Completion 2016-03 (Actual); Study Completion 2018-06-01 (Actual)

PRIMARY OUTCOMES:
recurrence of ankle sprain | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- MUHC-Montreal Children's Hospital, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No